CLINICAL TRIAL: NCT07106957
Title: A Single-center, Randomized, Double-blind, Controlled Study Lasting for 56 Days to Evaluate the Safety and Efficacy of LA ROCHE-POSAY CICAPLAST BAUME B5+ in Individuals With Rosacea Accompanied by Sensitive Skin
Brief Title: Efficacy and Safety Evaluation of CICAPLAST BAUME B5+ on Rosacea Accompanied by Sensitive Skin
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sino-German Union Cosmetic Institute Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025-033-YJ-012
Record Dates: First submitted 2025-07-14; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Erythematous Telangiectatic Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LA ROCHE-POSAY CICAPLAST BAUME B5+ (Experimental): During the first phase, after washing the face, the CICAPLAST BAUME B5+ group applies CICAPLAST BAUME B5+ on the whole face twice a day (morning and evening). During the second phase, after washing the face, both the CICAPLAST BAUME B5+ group and the standard cream group apply CICAPLAST BAUME B5+ on the whole face twice a day (morning and evening).
  Interventions: Other: CICAPLAST BAUME B5+
- Standard cream (Placebo Comparator): During the first phase,after wash face,Standard cream group apply the standard cream on whole face twice a day(morning and evening).During the second phase,after wash face, CICAPLAST BAUME B5+ group and standard cream apply the CICAPLAST BAUME B5+ on whole face twice a day(morning and evening).
  Interventions: Other: Standard cream

INTERVENTIONS:
Other: CICAPLAST BAUME B5+ — Twice a day (morning and evening) on face
  Arms: LA ROCHE-POSAY CICAPLAST BAUME B5+
Other: Standard cream — Twice a day (morning and evening) on face
  Arms: Standard cream

SUMMARY:
In total, 72 eligible research participants were recruited in this 56-day study. The participants were divided into two groups-namely the Experimental Group and the Control Group-according to stratified randomization, with 36 participants in each group. Finally, 30 participants in each group were expected to complete the study.

In this study, for patients with rosacea accompanied by sensitive skin, differences in repairing effects and other improvements were evaluated after they used LA ROCHE-POSAY CICAPLAST BAUME B5+ and a standard cream for 28 days, as well as differences between the two groups after both groups used LA ROCHE-POSAY CICAPLAST BAUME B5+ for an additional 28 days-via objective instrumental measurements and subjective assessments. Additionally, the safety of the investigational product was evaluated among these individuals.

DETAILED DESCRIPTION:
During the first phase, both the Experimental Group and the Control Group cleanse their face in the morning and evening according to their daily habits, and should maintain their usual cleansing method, product brand, dosage, etc. The Experimental Group uses the investigational product on the whole face (twice a day), while the Control Group uses the placebo product on the whole face (twice a day). Both groups use standard sunscreen in the morning. During the second phase, both groups use the investigational product on the whole face (twice a day) after cleansing according to their daily habits in the morning and evening, and use standard sunscreen in the morning. During the entire test period, research participants are not allowed to use any other facial skin care products except the provided investigational product or placebo, and the standard sunscreen.

The measurements will include clinical grading by dermatologists at Baseline (Day 0), Day 14 (after 14 days of application), Day 28 (after 28 days of application), Day 56 (after 56 days of application); Corneometer, Tewameter, pH meter, Chromameter, PeriCam PSI NR, VISIA; and self-grading at Baseline (Day 0), Day 14, Day 28, Day 56. Self-assessment will be conducted at Day0min (immediately after application), Day 14, Day 28, and Day 56. The 10% lactic acid stinging response test will be measured at Baseline (Day 0) and Day 28.

ELIGIBILITY:
Inclusion Criteria

* 18-55 years old
* Participants in the rosacea erythematous telangiectasia study or participants in the rosacea erythematous telangiectasia study who have not received treatment or have received treatment but are currently in a stable state (no treatment required). The treatment includes local medication, oral medication, phototherapy, or combined therapy
* The score of the Persistent Erythema Assessment Scale (CEA) is between 1 and 3 points
* The score of the Global Assessment Scale (IGA) is ≤2 points
* Dry facial skin
* People with sensitive skin (10% of those sensitive to lactic acid stinging)

Exclusion Criteria

* Intending to get pregnant, pregnant, lactating or within 6 months of delivery
* Research participants with other facial skin diseases (such as seborrheic dermatitis, systemic lupus erythematosus, facial miliform lupus, contact dermatitis, hormone-dependent dermatitis, etc.)
* Systemic diseases accompanied by severe organ damage, malignant tumors, chronic diseases with unstable control, acute infectious diseases, major surgeries or traumas, psychological and mental disorders, or other diseases that require local or systemic use of drugs or treatments that have an impact on acne
* The test area is accompanied by other skin diseases (dermatitis, eczema, infection, tumor, etc.) or has other skin conditions that interfere with evaluation (birthmarks, scars, etc.)
* Received physical, chemical or laser cosmetic surgery that is not for rosacea treatment within 3 months
* Subject who has participated in any clinical test during the past 2 month
* Others whose participation in the study is determined inappropriate by the dermatologist

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-08-10 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Corneometer | Baseline(Day 0), Day 14, Day 28, Day 56
  Skin hydration.The increase of Corneometer value indicates improvement of water content of skin.
Tewameter | Baseline(Day 0), Day 14, Day 28, Day 56
  Transepidermal water loss test. The lower value of TEWL indicates the better skin barrier function.
Chromameter | Baseline(Day 0), Day 14, Day 28, Day 56
  a* value. the smaller the value,the less red the skin .
pH meter | Baseline(Day 0), Day 14, Day 28, Day 56
  Skin pH level
Clinical grading-Clinician's Erythema Assessment | Baseline(Day 0), Day 14, Day 28, Day 56
  Clinician's Erythema Assessment(CEA).Score from 0 to 4( 0= Smooth;
  1= almost smooth;2= Mild;3= Moderate;4= Severe).The smaller the score value, the better.
Clinical grading-Investigator Global Assessment | Baseline(Day 0), Day 14, Day 28, Day 56
  Investigator Global Assessment(IGA).Score from 0 to 4( 0= Smooth;
  1= almost smooth;2= Mild;3= Moderate;4= Severe).The smaller the score value is, the better.

SECONDARY OUTCOMES:
Clinical grading-Visual Analogue Scale | Baseline(Day 0), Day 14, Day 28, Day 56
  Visual Analogue Scale(VAS).Skin dryness(Not dry at all 0- Very dry10),Burning(No burning sensation at all 0- Very burning 10),Stinging(No stinging sensation at all 0- Very stinging 10),Itching(No itching sensation at all 0- Very itching 10) ,Skin tightness(Not tight at all 0- Very tight 10).The smaller the score value, the better.
Clinical grading-Safety grading | Baseline(Day 0), Day 14, Day 28, Day 56
  Safety grading (Scaling, Congestion, Swelling, Blister, Infection, Exudation, Pigmentation, Hypopigmentation, Scar,other), The scale are: 0-None, 1-Very mild,2-Mild, 3-Moderate, 4-Severe.If the symptoms worsen, it is necessary to determine whether they are related to the product
Image analysis | Baseline(Day 0), Day 14, Day 28, Day 56
  VISIA 7 photos（a* value,Red area/AOI area[%]）. a* value,Red area/AOI area[%], the smaller the value,the less red the skin
PeriCam PSI NR | Baseline(Day 0), Day 14, Day 28, Day 56
  Blood perfusion volume.The higher the degree of blurriness, the greater the amount of blood flow attention; the lower the degree of blurriness, the smaller the amount of blood flow perfusion
Self-assessment | Immediately after once application(Timm),Day 14, Day 28, Day 56
  Self-assessment by subjects on face.The more percentages of "Full agree" & "Agree"are chosen, the better.
Self grading-Global Flushing Severity Score | Baseline(Day 0), Day 14, Day 28, Day 56
  Global Flushing Severity Score(GFSS).The smaller the score value, the better.
Self grading-Patient's Self-assessment Scale | Baseline(Day 0), Day 14, Day 28, Day 56
  Patient's Self-assessment Scale(PSA).The smaller the score value, the better. Score from 0 to 4( 0= Smooth;
  1= almost smooth;2= Mild;3= Moderate;4= Severe).The smaller the score value, the better.
Self grading-Rosacea-specific quality of life | Baseline(Day 0), Day 14, Day 28, Day 56
  Rosacea-specific quality of life(Rosa QOL).The smaller the total score, the better
Self grading-Dermatology Life Quality Index | Baseline(Day 0), Day 14, Day 28, Day 56
  Dermatology Life Quality Index(DLQI).The smaller the total score, the better
Self grading-The Sensitive Scale 14 | Baseline(Day 0), Day 14, Day 28, Day 56
  The Sensitive Scale 14(SS14),The smaller the total score, the better

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Sino-German Union Cosmetic Institute Co., Ltd., Beijing, China